CLINICAL TRIAL: NCT00000361
Title: Autoimmunity in Inner Ear Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDCD-1158; U01DC003209 (NIH)
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2006-04-24 (Estimated); Status verified 2006-04

CONDITIONS: Hearing Loss, Sensorineural
Keywords: Autoimmune Diseases; Cyclophosphamide; Hearing; Labyrinth Diseases; Methotrexate; Prednisone
MeSH Terms: conditions — Hearing Loss, Sensorineural; Autoimmune Diseases; Labyrinth Diseases | interventions — Adrenal Cortex Hormones; Methotrexate

INTERVENTIONS:
Drug: Corticosteroids
Drug: Methotrexate

SUMMARY:
The purpose of this study is to determine whether prednisone, methotrexate, and cyclophosphamide are effective in the treatment of rapidly progressive sensorineural hearing loss in both ears. This condition is called autoimmune inner ear disease (AIED), because it is thought that the hearing loss is triggered by an autoimmune process. Treatment attempts to suppress or control this process with powerful anti-inflammatory drugs. This is a Phase III, outpatient study. All study participants will be assigned to one of four different groups testing the experimental use of drugs. The study is scheduled to run for 18 months, with a minimum of 11 visits per participant.

ELIGIBILITY:
Inclusion Criteria:

* Have sensorineural (nerve/inner ear) hearing loss of at least 30 dB in each ear, which has rapidly progressed.
* Are in good general health.
* Are sterile or use contraception (if a woman of child-bearing age).
* Are able to speak and understand English or Spanish.

Exclusion Criteria:

* Have had any previous reaction to prednisone, or history of psychiatric reaction to corticosteroids.
* Have used corticosteroids for more than 30 days within the past 90 days. Patients who have been off corticosteroids for at least 30 days may be eligible.
* Have any significant heart, lung, digestive, blood, or neurologic disorders.
* Have tuberculosis (TB), brittle or unstable insulin-dependent diabetes mellitus, active malignancy or prior chemotherapy, pancreatitis, active peptic ulcer disease, kidney failure, history of shingles, or known (other) autoimmune disease.
* Have had a positive test for HIV, hepatitis C or B.
* Have any type of middle ear disorder.
* Are breast-feeding or pregnant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-03; Study Completion 2002-11

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Jeffrey Harris, Study Chair; Dr. Patrick Brookhouser, Principal Investigator
Locations (9):
- United States (9):
  - House Ear Institute, Los Angeles, California
  - UCSD Medical Center, San Diego, California
  - Univ of Iowa Hosp and Clinic, Iowa City, Iowa
  - Johns Hopkins Univ, Baltimore, Maryland
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - Univ of Michigan, Ann Arbor, Michigan
  - New York University, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Texas, Southwestern Medical Center at Dallas, Dallas, Texas